CLINICAL TRIAL: NCT05074927
Title: Pulmonary Function in Patients Recovering From COVID19 Infection : a Pilot Study
Acronym: EFRUPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 87RI20_0073
Record Dates: First submitted 2021-09-30; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: Lung function; Diaphragm ultrasonography; Chronic Inflammatory Rheumatism
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): All patients with confirmed COVID-19 who had been discharged from CHRU Hospital in Limoges (France)
  Interventions: Diagnostic Test: diaphragm ultrasonography

INTERVENTIONS:
Diagnostic Test: diaphragm ultrasonography — For all patients with confirmed COVID-19 who had been discharged from CHRU Hospital in Limoges (France) : diaphragm ultrasonography at 3 (M0) and 6 months (M3) after the end of his hospitalisation

SUMMARY:
The current state of knowledge shows the presence of respiratory sequelae after acute infection with COVID-19 and the importance of these long-term respiratory dysfunctions have to be determined.

Aim of our study is describe diaphragmatic amplitude using diaphragm ultrasonography in patients recovering from SARS-CoV-2 pneumonia at 3 and 6 months after the acute episode.

DETAILED DESCRIPTION:
patients with confirmed COVID-19 who had been discharged from CHRU Hospital in Limoges (France) will be included to follow the impact of severe acute respiratory syndrom coronavirus 2 on pulmonary function, diaphragm function and exercice capacity. Surviving patients will be evaluated at 3 and 6 months after hospital discharge. The assesment will include diaphragm ultrasonography, spirometry (FEV1,FVC), carbon monoxide transfert (TLCO adjusted for haemoglobin), inspiratory an expiratory respiratory muscle strength (Pimax and Pemax) and 6 minutes walk distance (6MWD).The main outcome will be diaphragm excursion assessed by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection proven by RT-PCR.
* Patient hospitalised for the management of SARS-CoV-2 infection and included 3 months after the end of his hospitalisation at the CHU of Limoges.
* Patient of legal age.
* Patient affiliated to a social security regime.
* Patient having given informed consent

Exclusion Criteria:

* Known pregnancy.
* Patients who are contraindicated to perform the 6-minute walk test.
* Patients unable to understand or adhere to the protocol.
* Patients deprived of liberty.
* Patients under court order, tutorship or curatorship.
* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
The change diaphragmatic amplitude using diaphragm ultrasonography in patients recovering from SARS-CoV-2 pneumonia. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  Diaphragmatic amplitude assessed by ultrasound at M0 and M3.

SECONDARY OUTCOMES:
the correlation between the values of diaphragmatic travel and Pi max and Pe max at M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  Diaphragmatic amplitude, PI max and PE max
the difference in diaphragmatic amplitude between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  Diaphragmatic amplitude at M0 and M3
the difference in FEV1 between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  FEV1 at M0 and M3.
the difference in FVC between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  FVC at M0 and M3.
the difference in DLCO between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  DLCO at M0 and M3.
the difference in Pi max and Pe max between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  PI max and PE max at M0 and M3
dyspnoea between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  mMRC dyspnoea scale at M0 and M3.
the functional capacity between M0 and M3. | at 3 (M0) and 6 months (M3) after the end of his hospitalisation at the CHU of Limoges
  6-minutes walk test distance at M0 and M3.

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT François, Pr, Principal Investigator — CHU Limoges